CLINICAL TRIAL: NCT06711484
Title: Evaluation of The Effıciency Of Speaking Up Training Program Developed For Newly Graduate Nurses
Brief Title: Evaluation of the Efficiency of a Training Program Developed For Newly Graduate Nurses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurcan Çalışkan, Professor of Nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-946; 2024-9261 (Other Grant/Funding Number: GAZİ ÜNİVERSİTESİ ARAŞTIRMA PROJELERİ BİRİMİ (BAP))
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Patient Safety; Nurse Training; Communication
Keywords: patient safety; newly graduated nurses; Speaking-Up; training program; transition shock; empowerment
MeSH Terms: conditions — Communication; Empowerment

STUDY DESIGN:
Intervention Model Description: This research is a randomized, pretest-posttest control group, parallel group experimental study that will evaluate the effectiveness of the language training program developed for newly graduated nurses. An introductory information form and a pretest evaluation of the scales will be applied to the participants who accept to participate in the research seven days before the application. Then, the groups will be randomized by an expert other than the researcher and assigned to their groups. The language training program will be applied to the experimental group seven days after the pretest evaluations. No intervention will be made to the control group. The final evaluation of the scales will be made to both groups seven days after the experimental group participants complete the training program. The language training program evaluation form will also be applied to the experimental group participants and their opinions about the training program will be obtained.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the training will be provided by the researcher, blinding the researcher will not be possible.
  All participants in the intervention and control groups will think that they will receive the entire language training. It will be explained that the trainings will be planned on different dates, notifications will be sent to mobile phones regarding the start and end times of the trainings, and the nurse whose turn it is will be called to the training. In this way, blinding of the participant will be ensured.
  After the explanation, the same informed consent form will be signed by the intervention and control group nurses.
  The statistician will perform the statistical analyses without knowing which group is the intervention and which group is the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPEAKİNG UP TRAİNİNG GROUP (Experimental): A pre-test will be administered to all participants seven days before the training program begins. A language training program consisting of four modules will be given to the experimental group participants. The final test of the scales and the training program evaluation form will be administered to the experimental group participants seven days after the training program is completed.
  Interventions: Other: Speak up traning program
- NON-TRAİNİNG GROUP (No Intervention): A pre-test will be applied to all participants seven days before the training program begins. No intervention will be made to the control group participants. The post-test of the scales will be applied to the control group again seven days after the training program of the experimental group participants is completed.

INTERVENTIONS:
Other: Speak up traning program — The intervention includes the training program to be applied to the experimental group. The aims and objectives of the training program, the training content and modules were prepared by the researcher in line with the needs analysis. The training program consists of four modules: Communication, Speaking UP, Patient Safety and Medical Error. Before the training program starts, the training booklet will be distributed to the experimental group participants. In the training, teaching techniques such as plain narration, question and answer, brainstorming, case study, case discussion, station technique, six thinking hats technique, video-based error scenario activity etc. will be used. The video activity to be used in the speak up session of the training program was created by recording the correct and incorrect scenarios of three patient safety errors by experienced actors.
  Arms: SPEAKİNG UP TRAİNİNG GROUP

SUMMARY:
Brief Summary: This research is a randomized, pre-test post-test control group, parallel group experimental study to evaluate the effectiveness of the language training program developed for newly graduated nurses. The study will be conducted with a total of 76 newly graduated nurses, 38 in the experimental group and 38 in the control group, at Etlik City Hospital Orthopedics-Neurology Hospital in Ankara. Participants will be informed about the study at the beginning of the study. Participants who agree to participate in the study and meet the eligibility criteria will be randomly assigned to groups by an independent statistician. The language training program will be applied to the experimental group, while no intervention will be made to the control group. The training program to be given to the experimental group will consist of a total of two days and four sessions (communication, speaking, patient safety, medical error), and each session will last 90 minutes. Data collection forms will be applied to the experimental and control groups before and after the training. Data collection forms include the descriptive characteristics form, working voice scale, effective communication skills scale, attitude scale in medical errors, and feedback about the language training program. Blinding of the raters will be applied to the participants to minimize bias. Data analysis will use statistical software that uses parametric tests for normally distributed data and nonparametric tests for non-normally distributed data.

DETAILED DESCRIPTION:
Purpose of the Study

The purpose of the study is to evaluate the effectiveness of the speak-up training program developed for newly graduated nurses.

Hypotheses of the Study H0-1: The speak-up training program has no effect on the employee voice levels of newly graduated nurses.

H1-1: The speak-up training program has an effect on the employee voice levels of newly graduated nurses.

H0-2: The speak-up training program has no effect on the effective communication skill levels of newly graduated nurses.

H1-2: The speak-up training program has an effect on the effective communication skill levels of newly graduated nurses.

H0-3: The speak-up training program has no effect on the medical error attitude levels of newly graduated nurses.

H1-3: The speak-up training program has an effect on the medical error attitude levels of newly graduated nurses.

Variables of the Study

Independent variables

• Socio-demographic characteristics of the new graduate nurses

Dependent variables

* Total score of the Employee Voice scale after the implementation of the training program developed for the speaking up of new graduate nurses
* Total and sub-dimension scores of the Communication Skills scale after the implementation of the training program developed for the speaking up of new graduate nurses Total and sub-dimension scores of the Attitude to Medical Errors scale after the implementation of the training program developed for the speaking up of new graduate nurses
* Evaluations of the training program developed for the lspeaking up of new graduate nurses

Population and Sample of the Study

The population of the study will consist of 152 newly graduated nurses working at Etlik City Hospital Campus Orthopedics-Neurology Hospital. The characteristics of the newly graduated nurses selected for this study are that they have completed basic nursing professional education, have been in the clinic for the first two years after graduation, and have not received speaking up training. The sample size of the study was determined by power analysis (G*Power 3.1 program). In a similar study in the relevant literature, in the study conducted by Walther et al. (2022), the effect size for the difference in vocalization between the groups (Effect size) was 0.811. In order to exceed the 95% value in determining the power of the study; 68 people, 34 in the groups, should be reached at a significance level of 5% and an effect size of 0.811 (df=66; t=1.668). Considering the high power of the test and the losses in the study, a total of 76 people, 38 in the groups, will be reached.

Randomization: Randomization will be performed by a doctoral education nurse at the institution where the researcher, who is not involved in the study, works. The researcher will not intervene in the randomization list. Newly graduated nurses who meet the inclusion criteria and agree to participate in the study will be assigned to the intervention and control groups. Impartiality will be ensured by the random assignment of the intervention and control groups.

Blinding:

Since the patient safety language training will be provided by the researcher in the study, blinding the researcher will not be possible.

In order to blind the participants, all nurses in the intervention and control groups will think that they will receive the entire language training. It will be explained that the tests and trainings to be conducted regarding the study will be planned on different dates, notifications will be sent to mobile phones regarding the start and end times of the trainings, and the nurse whose turn it is will be called to the training. After the explanation, the same informed consent form will be signed by the intervention and control group nurses.

The statistician will perform the statistical analyses without knowing which group is the intervention and which group is the control. The randomization process was carried out in accordance with the CONSORT 2017 guidelines.

Descriptive Characteristics Form The Descriptive Characteristics Form consists of seven questions that will determine individual information such as nurses' age, gender, education level, unit they work in, working hours, and working style. In addition, the form will include two questions to determine nurses' views on voicing.

Employee Voice Scale Van Dyne and LePine (1998) developed the employee voice scale as a 6-item, single-dimensional scale. In our country, the Employee Voice Scale was adapted to Turkish by Çetin and Çakmakçı (2012). All items in the scale are measured according to a 5-point Likert scale. Higher scores indicate more employee voice behavior.

Effective Communication Skills Scale The Effective Communication Skills Scale consists of 5 sub-dimensions and a total of 34 items and was developed by Buluş et al. (2017). Items 15, 16, 28, 32 and 33 of the scale are scored reversely. Therefore, as the total score obtained from each sub-dimension increases, the level of using communication skills also increases.

Attitude Scale on Medical Errors The scale was developed by Güleç and İntepeler in 2012 and consists of three sub-dimensions, namely perception of medical error, approach to medical error and causes of medical errors, and 16 questions. The scale is a five-point Likert type. If the average score obtained from the scale is 3, it indicates that attitudes towards medical errors are negative, and if it is 3 and above, it indicates that attitudes towards medical errors are positive.

Evaluation Form for the Speak-up Training Program

Araştırmacı literatürü takip ederek dil eğitimlerinin birleştirilmesini sağlamak amacıyla hazırlandı. Bu form iki bölümden oluşur. Literatür taramasına dayalı birinci bölüm, eğitim programı içeriği, eğitim süresi, kullanılan öğretim bölümleri, değerlendirme yöntemi ve eğitimin algılanan etkililiği olmak üzere toplam 16 maddeden oluşmaktadır. İkinci bölüm, dil eğitim programları teorik ve video içeriği hakkında yayınlama soran dört açık uçlu sorudan oluşmaktadır.

İçerik Rekabetçilik Analizi İçerik bakımı, iletişim, hasta güvenliği, dil ve eğitim alanlarında 7 uzmana danışılarak değerlendirilmiştir. Formları amaç, hedefler, dil ve anlam açısından 4 puanlık Likert performansında derecelendirildiler (4: Çok uygun, 3: Küçük ayarlamalarla uygun, 2: Büyük ayarlamalarla uygun, 1: Uygun değil). Uzman yayın, içerik düzenliliği programlaması için Davis teknolojisi kullanılarak analiz edilmiştir.

Development of Speak-up Training Program

The language training program was developed using the ADDIE model. The model consists of analysis, design, development, implementation and evaluation stages.

The language training program was developed using the ADDIE model. The model consists of analysis, design, development, implementation and evaluation stages.

Analysis

The researcher conducted a nine-question interview with manager nurses, education and quality unit nurses, infection control nurses, hemovigilance nurses, responsible nurses and experienced nurses working at Etlik City Hospital and participating in the study voluntarily to determine the needs of the participants regarding the language training program. The researcher analyzed the characteristics, experiences and work environments of the participants and reviewed the hospital adverse event notification reports. The literature review was conducted as a retrospective review of publications to determine the content, learning objectives and learning areas of the training program. For this purpose, the keywords speak up, nurses, nursing, education, (training), intervention, program, curriculum, guide were used in the Turkish and English title and abstract fields from the Pubmed (29), Cohrane (4), Google Academy (33), Medline (38), Science Direct (12) databases between 2018-2023.

Design

The researcher determined the measurement and evaluation tools to be used in the study. Developed a language education program evaluation form. Created theoretical education contents, language video scenarios and video discussion questions.

Development

The content of the training program, the materials used, the measurement and evaluation tool and the scenarios were reviewed by the experts. The researcher made adjustments based on the feedback. The professional actors were informed about the scenario and the training video was shot. The researcher made a preliminary application of the training program and made the necessary corrections

Implementation

The implementation phase of the study includes the Implementation and Evaluation steps of the ADDIE design model.

Participants who will participate in the study will be informed about the training program, and the introductory information form and scales will be applied. Then, participants will be randomly selected and assigned to the research groups. One week after the completion of the pre-test applications, the implementation of the language training program for the experimental group will begin. In order to ensure effective and easy participation of the participants in the training, the "Speaking Up Training Program" trainings will be held in the Orthopedics-Neurology Hospital training class. Before the start of the training program, the training booklet containing advanced reading resources and training contents will be distributed to the experimental group participants. The language training program will consist of four sessions and each session will last 90 minutes.

Seven days after the completion of the training program, the final evaluation of the scales will be made to the experimental and control group nurses.

Analysis:

The data will be analyzed using a computer program. The normal distribution of variables will be evaluated with histogram, coefficient of variation, skewness, kurtosis, Kolmogorov-Smirnov and Shapiro-Wilk tests (p<0.05). Descriptive statistics (number, percentage, mean, standard deviation) and Chi-square tests will be used. Parametric tests will be applied to data showing normal distribution, and nonparametric tests will be applied to data not showing normal distribution. Independent sample t-test will be used for comparisons between two independent groups, ANOVA with Bonferroni correction for comparisons between two or more groups, and variance analysis for repeated measurements. Mann-Whitney U and Kruskal-Wallis H tests with Bonferroni correction will be applied for data not showing normal distribution. Randomization balance will be provided using Intention to Treat (ITT) analysis.

Limitations

A limitation of this study is that only new graduate nurses working in one hospital and who agreed to participate in the study were included in the study. The results cannot be generalized to all new graduate nurses.

The fact that the gender and professional experience characteristics of the newly graduated nurses included in the study were concentrated on one side limited the use of stratified block randomization.

ELIGIBILITY:
Inclusion Criteria:

* Having a maximum of two years of post-graduation professional experience
* Having a minimum of three months of post-graduation professional experience
* Being willing to participate in the research
* Having completed general orientation training

Exclusion Criteria:

* Having received previous training in language translation
* Those with education below undergraduate level

Exclusion criteria for the study:

* Not having attended the entire training program
* Not having completed all the data collection tools
* Wanting to leave the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
Employee Voice Scale | It will be evaluated seven days before the intervention (pre-test) and seven days after the intervention (post-test).
  The Employee Voice Scale was developed by Van Dyne and LePine and is a 6-item, single-dimensional scale. In our country, the Employee Voice Scale was adapted to Turkish by Çetin and Çakmakçı. All items in the scale are measured on a 5-point Likert-type scale using the following scales: disagree, somewhat agree, partially agree, mostly agree, completely agree. Higher scores indicate more employee voice behavior.

SECONDARY OUTCOMES:
Effective Communication Skills Scale | It will be evaluated seven days before the intervention (pre-test) and seven days after the intervention (post-test).
  The Effective Communication Skills Scale consists of 5 sub-dimensions and a total of 34 items. The scale consists of the sub-dimensions "ego-enhancing language" (6 items), "active listening" (8 items), "self-awareness/self-disclosure" (5 items), "empathy" (8 items) and "I language" (7 items). As the total score from each sub-dimension of the scale increases, the level of using communication skills also increases.
Attitude Scale in Medical Errors | It will be evaluated seven days before the intervention (pre-test) and seven days after the intervention (post-test).
  The scale was developed by Güleç and İntepeler and consists of three sub-dimensions, namely perception of medical error, approach to medical error and reasons for medical error, and 16 questions. The scale is a five-point Likert type. The items are Strongly disagree, Disagree, Undecided, Agree and Strongly agree. The total score of the scale varies between 1-5. The average score obtained from the scale is 3, indicating that attitudes towards medical errors are negative, and a score of 3 and above indicates that attitudes towards medical errors are positive.
Evaluation Form for the Speaking-Up Training Program | It will be collected immediately after the intervention.
  The researcher prepared the form by following the relevant literature in order to measure the opinions on the language education program. This form consists of two parts. The first part, based on the literature review, consists of a total of 16 items, including the content of the education program, duration of education, teaching materials used, evaluation method and perceived effectiveness of education. The second part consists of four open-ended questions asking opinions on the theoretical and video content of the language education program.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Nursing Faculty, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akın, B. ve Koçoğlu, D. Randomize Kontrollü Deneyler. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi. 2017 4(1): 73-92.
- [Background] Van Dyne, L. ve LePine, J.A. (1998). Helping and voice extra-role behavior: Evidence of construct and predictive validity. Academy of Management Journal, 41, 108-119.
- [Background] Çetin, Ş. ve Çakmakçı, C. (2012). Çalışan Sesliliği Ölçeğini Türkçeye Uyarlama Çalışması. Kara Harp Okulu Bilim Dergisi, 22(2), 1.
- [Background] Güleç, D. ve İntepeler, Ş.S. (2013). Tıbbi hatalarda tutum ölçeğinin geliştirilmesi. Hemşirelikte Araştırma Geliştirme Dergisi, 15:3, 26-41.
- [Background] Buluş, M., Atan, A., & Sarıkaya, H. E. (2017). Effective Communication Skills: A New Concep-tual Framework and Scale Development Study. International Online Journal of Educational Sci-ences, 9(2).
- [Background] Lee SE, Kim E, Lee JY, Morse BL. Assertiveness educational interventions for nursing students and nurses: A systematic review. Nurse Educ Today. 2023 Jan;120:105655. doi: 10.1016/j.nedt.2022.105655. Epub 2022 Nov 25. PMID 36462396
- [Background] Wawersik DM, Boutin ER Jr, Gore T, Palaganas JC. Individual Characteristics That Promote or Prevent Psychological Safety and Error Reporting in Healthcare: A Systematic Review. J Healthc Leadersh. 2023 Apr 17;15:59-70. doi: 10.2147/JHL.S369242. eCollection 2023. PMID 37091553
- [Background] Lee SE, Choi J, Lee H, Sang S, Lee H, Hong HC. Factors Influencing Nurses' Willingness to Speak Up Regarding Patient Safety in East Asia: A Systematic Review. Risk Manag Healthc Policy. 2021 Mar 12;14:1053-1063. doi: 10.2147/RMHP.S297349. eCollection 2021. PMID 33737846
- [Background] Lee E, De Gagne JC, Randall PS, Kim H, Tuttle B. Effectiveness of speak-up training programs for clinical nurses: A scoping review. Int J Nurs Stud. 2022 Dec;136:104375. doi: 10.1016/j.ijnurstu.2022.104375. Epub 2022 Oct 7. PMID 36327680
- [Background] O'Donovan R, McAuliffe E. A systematic review exploring the content and outcomes of interventions to improve psychological safety, speaking up and voice behaviour. BMC Health Serv Res. 2020 Feb 10;20(1):101. doi: 10.1186/s12913-020-4931-2. PMID 32041595